CLINICAL TRIAL: NCT04866693
Title: Understanding the Nature of the Safety and Quality of Care Problems Experienced by Service Users Accessing Community-based Mental Health Services: a Qualitative Study
Brief Title: Improving Safety and Quality in Mental Healthcare
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 279409
Record Dates: First submitted 2021-04-22; First posted 2021-04-30 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Mental Illness
Keywords: Patient safety; Community mental health services
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Service users: Up to 20 people with current or recent experience of using community-based mental health services will be recruited to the study. Participants will take part in one in-depth interview or focus group discussion.
  Interventions: Other: None - this is an exploratory qualitative study to understand patient safety problems in community-based mental healthcare.
- Carers: Up to 20 family members/ carers with experience of supporting another adult who is accessing community-based mental health services, will be recruited to the study. Participants will take part in one in-depth interview or focus group discussion.
  Interventions: Other: None - this is an exploratory qualitative study to understand patient safety problems in community-based mental healthcare.
- Healthcare professionals: Up to 20 healthcare professionals from different disciplinary backgrounds and community-based mental health services will be recruited to the study. Participants will take part in one in-depth interview or focus group discussion.
  Interventions: Other: None - this is an exploratory qualitative study to understand patient safety problems in community-based mental healthcare.

INTERVENTIONS:
Other: None - this is an exploratory qualitative study to understand patient safety problems in community-based mental healthcare. — Qualitative study

SUMMARY:
Background:

Patient safety incidents are a leading cause of death and disability worldwide. So far, existing safety improvement work has largely focused on physical healthcare. Only a small body of research has studied safety as it applies to mental healthcare, with these studies concentrating primarily on psychiatric inpatient units. However, mental healthcare is increasingly delivered in community settings, through primary care and secondary care mental health provision, rather than in hospitals. Less is known about the safety problems service users experience in community-based mental healthcare. It is important that safety problems in community-based mental health services are better understood, so that care can be improved.

Objective:

This research will aim to understand the nature of the safety problems experienced by adult users of community-based mental healthcare, from the perspective of service users, carers, and healthcare providers. The study will also aim to identify priority areas and effective practices to improve safety in these settings.

Method:

Individual in-depth interviews or focus groups will be held with service users, carers, and frontline healthcare providers employed within appropriate community-based mental healthcare settings. Interviews or focus groups will last for approximately one hour and will be carried out face-to-face or via secure videoconferencing technology (e.g. Microsoft Teams or Zoom), depending on up-to-date guidance relating to the Covid-19 pandemic. With participant consent, interviews and focus groups will be audio-recorded and transcribed. Transcripts will be analysed using thematic analysis, with themes developed, defined, and revised throughout the analysis process.

Discussion:

Study findings will help to fill key evidence gaps concerning safety in community-based mental healthcare. More broadly, the results may lead to the development of evidence-informed interventions to address the safety issues which are raised in participant discussions.

DETAILED DESCRIPTION:
Background:

Patient safety problems are widespread. Research suggests that around 10% of inpatients experience an adverse event during their hospital admission, with almost half of these incidents judged to be preventable. There have been considerable advancements in initiatives to improve patient safety in medical settings in the past 20 years. However, safety in mental healthcare remains an under-researched and poorly understood issue, with only a limited amount of research having explored safety as it uniquely applies to this population. Self-harm, suicide, and coercive interventions (such as physical restraint) are some of the specific risks which may affect mental health service users.

The small body of research focusing on safety in mental healthcare has primarily concentrated on hospital-based inpatient care. This is problematic for improving mental healthcare safety and quality, as only a minority of mental healthcare episodes take place within psychiatric inpatient services. As such, research into the types of safety problem experienced by users of community-based mental healthcare is of great importance to improving care and reducing harm.

Despite a willingness to share their perspectives, mental health service users and carers have reported barriers to raising their safety concerns with professionals. These include feeling as if their concerns were not listened to, as well as challenges associated with the process of raising a complaint whilst unwell. Likewise, frontline care providers and service managers within mental health services can also provide different yet complementary professional insights into safety.

Community-based mental healthcare provision is diverse, often involving complex relationships between and joint responsibly of multiple agencies. Because of this, the safety problems associated with different care pathways are likely to be varied in nature. In order to fully understand safety and broader quality of care problems, it is important to draw upon the perspectives of mental health service users, carers, and healthcare providers from a range of community settings. Using qualitative research methods, this research will begin to address this evidence gap, focusing on services for working-aged adults.

Aims:

The primary aim of this study is to gain a deeper understanding of the safety problems which occur in the context of community-based mental healthcare. Specifically, drawing upon the perspectives of multiple stakeholder groups, including service users, carers and frontline care providers, the objectives are to investigate the following:

1. To explore perspectives on the meaning of 'safety' in mental healthcare;
2. To understand the nature of the safety problems faced by people accessing community-based mental health services;
3. To learn about experiences of good practice in the delivery of safe mental healthcare;
4. To identify priority areas and strategies for intervention to improve care safety.

Study design:

The study design will comprise in-depth qualitative interviews or focus groups, with three participant groups: (a) working-age adult service users, (b) carers, (c) staff within community-based mental health services (frontline providers and service managers). The research team consulted with service users and carers about the study design, and received positive feedback about the proposal to conduct either individual qualitative interviews or focus groups.

Data analysis:

Interviews and focus groups will be audio-recorded and transcribed verbatim by a professional transcription company from King's College London's list of approved suppliers. Prior to analysis, any interview or focus groups excerpts containing information which could potentially identify the participant, will be redacted. Interview and focus group data will be managed in NVivo and analysed using a reflexive approach to thematic analysis, according to the methodologies outlined by Braun and Clarke (2006). Themes will be developed and revised through an iterative process.

Paper consent forms will be stored in a locked filing cabinet within the university premises, to which only the research team will have access. Digital files, such as interview transcripts and electronically completed consent forms, will be stored on the researcher's secure university account server, which is password protected. Audio recordings will also be stored here up until the point of transcription, after which they will be securely deleted. Data will be stored anonymously and archived in line with King's College London's policy on data storage.

Study setting:

This study will focus on service users, carers, and staff members employed within general adult community-based mental health services. Community-based mental health services herein refers to non-institutional mental health services which deliver multidisciplinary care accessed by service users living independently, or in supported accommodation (excluding settings with 24-hour on-site care from qualified nurses, which resemble institutional care models). As such, participants associated with a range of settings may be recruited, including community mental health services within secondary care (e.g. Assertive Outreach Services) and mental health support available through primary care (e.g. from a general practitioner).

Sampling:

In order to capture a range of perspectives, participants will be purposively sampled according to several key characteristics. The recruitment strategy will aim to recruit service users, carers, and healthcare professionals who have experience of different types of community-based mental health services. To reflect the range of care contexts and professional roles, the investigators will seek to sample healthcare professionals from different disciplinary backgrounds. This will likely include clinical service managers, psychiatrists, occupational therapists, nurses, social workers, and psychologists. Efforts will be made to recruit people within each group who represent a range of sociodemographic characteristics, including participants of different sexes and from different ethnic groups.

Potential participants will be recruited via community-based mental health services and via an open recruitment call (e.g. via online advertisements, or existing service user and carer network newsletter mailings). Snowball sampling techniques may also be used to supplement the sample. As such, recruited participants may be asked to invite other people they know to contact the research team directly, if they are interested in taking part and meet the study eligibility criteria. These sampling approaches have been selected due to their appropriateness for qualitative research which seeks to capture the range and diversity of participant perspectives, rather than aiming to achieve a representative study sample.

Procedure:

Those who express interest in taking part will receive a participant information sheet at least 24 hours before taking part in a scheduled interview or focus group. Potential participants will have the opportunity to ask questions and receive further information about the study before deciding whether to take part and providing their informed consent. Interviews or focus groups will last for approximately one hour and be conducted in a private space. Interviews and focus groups will be primarily conducted remotely (due to COVID-19 safety considerations) via secure digital communications software (e.g. Microsoft Teams or Zoom). Where face-to-face interviews are held, these will be conducted in accordance with up-to-date safety guidance.

ELIGIBILITY:
Service users.

Inclusion criteria:

* Over 18 years old.
* Able to speak sufficient English to provide informed consent to take part in an interview or focus group.
* Current or prior experience of using general adult community-based mental health services (within the past 12 months).

Exclusion criteria:

* Unable to speak sufficient English to take part in an interview or focus group.
* Unable to give informed consent to take part in an interview or focus group.
* Currently receiving inpatient mental healthcare at a psychiatric hospital, or care from a service for older adults.
* Deemed by the researcher to be distressed or too unwell to take part in an interview or focus group.
* Their experience of services primarily falls outside of the remit of general adult mental health services, e.g. they have a primary diagnosis of Substance Use Disorder, or their care is provided by specialist tertiary care providers such as forensic mental health services.

Carers.

Inclusion criteria:

* Over 18 years old.
* Able to speak sufficient English to provide informed consent to take part in an interview or focus group.
* Current or prior experience of caring for an individual accessing general adult community-based mental health services (within the past 12 months).

Exclusion criteria:

* Unable to speak sufficient English to take part in an interview or focus group.
* Unable to give informed consent to take part in an interview or focus group.
* Carers who have a caring responsibility for:

  * A child (0-17 years),
  * An individual using older adult mental health services,
  * An adult using services which fall outside of the remit of general adult mental health services,
  * Someone without a mental health problem.

Healthcare professionals.

Inclusion criteria:

* Over 18 years old.
* Able to speak sufficient English to provide informed consent to take part in an interview or focus group.
* Currently employed within a community-based service which provides general adult mental healthcare.

Exclusion criteria:

* Unable to speak sufficient English to take part in an interview or focus group.
* Unable to give informed consent to take part in an interview or focus group.
* Healthcare professionals who are currently working in a mental health service which:

  * Is not based in a community setting (e.g. inpatient care),
  * Falls outside of the remit of general adult mental health services,
  * Provides services to children (0-17 years) or older adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with experience of community-based mental health services, in either a service user, carer, or healthcare professional capacity.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Safety problems in community-based mental health services | The outcome will be assessed on day 1 of participation, during a one-off interview/focus group
  In-depth qualitative interviews or focus group discussions will be conducted to identify patient safety problems within community-based mental health services, from the perspective of each participant group (service users, carers, healthcare professionals).

CONTACTS AND LOCATIONS:
Overall Officials: Claire Henderson, FRCPsych, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, King's College London, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04866693/ICF_000.pdf